CLINICAL TRIAL: NCT03302819
Title: Performance Evaluation of the MARIA (Multi Static Array Processing of Radiowave Image Acquisition) Radar Breast Imaging System in Patients With Breast Cancer and in Patients Assessed in the Symptomatic Breast Clinic.
Brief Title: London Investigation Into diElectric Scanning of Lesions
Acronym: LIESL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Micrima, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CCR4702
Record Dates: First submitted 2017-09-21; First posted 2017-10-05 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Breast cancer accuracy (Experimental): Patients with a known or suspected (and subsequently proven) breast cancer
  Interventions: Diagnostic Test: MARIA scan
- Imaging characteristics and performance (Experimental): Patients attending the symptomatic clinic
  Interventions: Diagnostic Test: MARIA scan
- Tumour response in neoadjuvant treatment (Experimental): Patients who are being treated with neoadjuvant chemotherapy or endocrine treatment
  Interventions: Diagnostic Test: MARIA scan

INTERVENTIONS:
Diagnostic Test: MARIA scan — The patient will have an additional MARIA scan along with conventional imaging, pathology and surgical procedures.

SUMMARY:
The MARIA breast imaging system is a novel CE-marked radio-frequency (RF) medical imaging device. The system employs an electromagnetic imaging technique that exploits the dielectric contrast between normal and cancerous tissues. The performance and imaging characteristics of MARIA are not yet well demonstrated. The investigators aim to evaluate some aspects of this potentially important new technology.

DETAILED DESCRIPTION:
The early diagnosis of breast cancer is of paramount importance, with a 5-year survival rate of 97% if the cancer is caught "locally", deteriorating to 79% if it has progressed to the "axillary" lymph nodes, and 23% if it has spread to the rest of the body, known as "metastasised."

Diagnosis is currently achieved through clinical examination, imaging with mammography (MMG) and/or ultrasound (US) and needle biopsy. Mammography is dependent upon adequate breast compression to allow greater contrast differentiation between tissue structures, this is not only uncomfortable, but in younger women with 'dense' breast tissue the contrast difference between normal tissue and tumour is minimal despite compression. Furthermore mammography uses ionising radiation, which means that a risk/benefit calculation is weighted against repeated or frequent use. Frequently it is necessary to use additional imaging such as ultrasound or MRI for diagnostic support.

Breast tumours have an additional property that can distinguish them from normal and this is defined by the dielectric value. This has two components - the dielectric constant, which affects the velocity of propagation of radio waves and therefore their wavelength, and the conductivity, which affects the rate of attenuation. Typically a tumour has a dielectric constant of 45-50 and a conductivity of 2S/m, whereas breast fat is 5-15 and 0.2-1S/m respectively but with considerable range. Normal glandular tissue is intermediate. These differences in dielectric constant enable a consideration of the value of this data in breast cancer diagnosis.

Several attempts to exploit this property for imaging have been made. The outcomes have been similar in that the presence of a tumour is detectable, however limitations in depth for detection and mode of the technology were identified.

Due to updated technology in the MARIA device, previous limitations from similar studies are not reported to be a problem.

This study aims to determine the proportion of patients with breast cancer who are correctly diagnosed by MARIA, and to stratify this by breast density and histological type. In addition a pilot study will be performed to investigate the imaging characteristics and performance of MARIA in the assessment of benign and malignant lesions in patients attending the symptomatic breast clinic.

The MARIA scan will be in addition to any standard diagnostic procedures, including imaging, that comprise the standard of care. The scan will require them to lie prone for less than 10 minutes with their breast pendant in an ergonomically-fitted bowl with a thin layer of a coupling fluid (similar to hand moisture in consistency) applied to the surface of the breast.

While there is no direct benefit nor detrimental effect from this study to the patients participating, the study has large implications for many women.

This study will allow the investigators to test the feasibility of this highly innovating approach to breast cancer, with minimal negative effects or possible complications. This diagnostic modality could prove to be a major step forwards in cancer detection, initially as a complementary source of information that can increase confidence in results obtained from established technologies that are routinely deployed in the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Attending a symptomatic breast care clinic OR Patients who have a diagnosed or suspected breast cancer (P5/M5/U5/B5).
* Female sex
* 18 years or older.
* Able to provide informed consent.
* Not in any identified, vulnerable group.

Exclusion Criteria:

* Unable to mount MARIA™ patient bed using provided 2-step
* Unable to lie in the prone position
* Patients who have undergone biopsy less than 5 days before the MARIA™ scan
* Patients with implanted electronics.
* Patients with breast implants.
* Patients with nipple piercings (unless they are removed prior to the MARIA™ scan)
* Breast sizes smaller than 197ml or greater than 1L in volume

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 994 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-11-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with breast cancer in whom breast cancer is correctly identified by MARIA | 1 week (after histopathology result)
  Comparison to histopathology result
Sensitivity and specificity of MARIA for a range of findings to include, simple cysts, fibroadenomata, and malignant lesions. As judged against the final diagnosis at discharge, which may be based on clinical findings, imaging and pathology data. | Through study completion, an average of 1 year
  Comparison with clinical, radiology and pathology findings
Proportion of post-operative patients treated with neo-adjuvant chemotherapy or endocrine therapy, correctly identified by MARIA with complete response or residual disease, as compared to surgical histology. | Through study completion, an average of 1 year
  Comparison of response to surgical histology

SECONDARY OUTCOMES:
Compare the detection of breast cancer from MARIA with the detection from mammography by the sub-group of histology type. | Through study completion, an average of 1 year
  Comparison to Mammography and Pathology result
Compare the detection of breast cancer from MARIA with the detection from mammography by sub-group of mammographic density. | Through study completion, an average of 1 year
  Comparison to Mammography and Pathology result
Compare the detection of breast cancer from MARIA with the detection from mammography in the overall patient group. | Through study completion, an average of 1 year
  Comparison to Mammography and Pathology result
Assessment of data repeatability (test re-test) of MARIA assessment results on patients with diagnostic follow-up imaging. | After attendance for further imaging, at 1-2 weeks.
  Comparison with prior MARIA scan when returning for further imaging
Investigate the performance of MARIA in the estimation of residual tumour size compared to the final surgical histology results in the case of patients receiving neo-adjuvant chemotherapy or endocrine therapy. | Through study completion, an average of 1 year
  The correlation between the pathological features of the lesion and the imaging features as determined from MARIA including presence of features, shape and size.
Patient tolerance of MARIA (a non-compressing, non-ionising modality) | Through study completion, an average of 1 year
  Questionnaire measurement, Quantitative answers.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Allen, Study Chair — Royal Marsden NHS Foundation Trust; Richard Sidebottom, Principal Investigator — Royal Marsden NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Preece AW, Craddock I, Shere M, Jones L, Winton HL. MARIA M4: clinical evaluation of a prototype ultrawideband radar scanner for breast cancer detection. J Med Imaging (Bellingham). 2016 Jul;3(3):033502. doi: 10.1117/1.JMI.3.3.033502. Epub 2016 Jul 20. PMID 27446970
- [Background] Saadatmand S, Bretveld R, Siesling S, Tilanus-Linthorst MM. Influence of tumour stage at breast cancer detection on survival in modern times: population based study in 173,797 patients. BMJ. 2015 Oct 6;351:h4901. doi: 10.1136/bmj.h4901. PMID 26442924